CLINICAL TRIAL: NCT06529003
Title: Randomized Controlled Trial: TENS Unit To Decrease Pain After Laminaria Insertion
Brief Title: TENS Unit To Decrease Pain After Laminaria Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's Medical Center (Other)
Collaborators: University of Hawaii Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RA-2024-018
Record Dates: First submitted 2024-07-09; First posted 2024-07-31 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Second Trimester Abortion
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Device: Placebo
- TENS unit (Active Comparator)
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS) unit

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation (TENS) unit — All participants in this study will receive the standard of care, which includes oral ibuprofen and a paracervical block at the time of laminaria insertion. Those in the treatment group will receive an adjunctive TENS unit with specific instructions for use in the interval between laminaria insertion and dilation and evacuation the next day. TENS is a non-invasive, inexpensive, over-the-counter, nonpharmacologic option to relieve pain. All participants will be provided with 15 tabs of ibuprofen 200 mg for outpatient pain control after the procedure. Participants will be instructed to take 600-800 mg of ibuprofen with food every 6 hours as needed for pain during the time period after laminaria insertion and before dilation and evacuation surgery, which is generally less than 24 hours.
  Arms: TENS unit
Device: Placebo — Participants in the placebo group will be given a TENS unit without a battery with similar to the intervention group but will be advised that they may or may not feel a sensation from the electrodes. All participants will be provided with 15 tabs of ibuprofen 200 mg for outpatient pain control after the procedure. Participants will be instructed to take 600-800 mg of ibuprofen with food every 6 hours as needed for pain during the time period after laminaria insertion and before dilation and evacuation surgery, which is generally less than 24 hours.
  Arms: Placebo

SUMMARY:
The purpose of the study is to learn more about the transcutaneous nerve stimulation (TENS) unit, an over-the-counter option for pain relief that is not a medication. The investigators are hoping to find out if this device decreases pain during and after laminaria placement for patients undergoing both elective and medically indicated second-trimester termination of pregnancy.

DETAILED DESCRIPTION:
To compare the maximum pain scores reported during the interval between osmotic dilator placement and D&E procedure of patients receiving the standard of care plus sham placebo and those who use an adjunctive Transcutaneous electrical nerve stimulation (TENS) unit in addition to standard of care.

Secondary objectives include comparing pain scores at the time of laminaria insertion, assessing the number and duration of TENS sessions, additional analgesic use, satisfaction with pain management, and patient perception of the ease of use of the TENS unit.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laminaria insertion for D&E procedure
* Age 18 years or older
* Capability and willingness to send and receive SMS messages by phone and complete web-based surveys
* Capability to read and understand directions for using a TENS unit
* Capability to operate a TENS unit according to provided directions

Exclusion Criteria:

* Inability to complete the informed consent in English
* Exposure to adjunctive pharmacologic cervical preparation (misoprostol or mifepristone) within 48 hours of the D&E procedure
* Contraindication to ibuprofen or bupivacaine
* Contraindication to TENS, including cardiac pacemakers, epilepsy, bleeding disorders, cancer, and concurrent use near transdermal drug delivery systems
* Previous participation in this trial
* Prior use of TENS unit

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-08-14 (Actual); Primary Completion 2025-11-05 (Actual); Study Completion 2025-11-05 (Actual)

PRIMARY OUTCOMES:
Maximum pain scores | Between osmotic dilator placement and dilation and evacuation procedure (approximately 16-24 hours)
  To compare the maximum pain scores reported during the interval between osmotic dilator placement and D&E procedure of patients receiving the standard of care plus placebo and those who use an adjunctive transcutaneous electrical nerve stimulation (TENS) unit in addition to standard of care. Participants will be asked to rank their pain on an 11-point numerical rating scale (0 to 10), with higher numbers indicating worse pain.

SECONDARY OUTCOMES:
Pain at time of laminaria insertion | At time of laminaria insertion
  Pain scores at the time of laminaria insertion. Participants will be asked to rank their pain on an 11-point numerical rating scale (0 to 10), with higher numbers indicating worse pain.
Number of TENS sessions | Between osmotic dilator placement and dilation and evacuation procedure (approximately 16-24 hours)
  Number of TENS sessions
Duration of each TENS sessions | Between osmotic dilator placement and dilation and evacuation procedure (approximately 16-24 hours)
  Duration of each TENS sessions
Satisfaction with pain management | Between osmotic dilator placement and dilation and evacuation procedure (approximately 16-24 hours)
  Participants will be asked "Overall satisfaction with pain control since the procedure: (0-10 numeric rating scale)" on all five surveys. A score of 0 indicates "extremely unsatisfied." A score of 5 indicates "neutral." A score of 10 indicates "extremely satisfied."
Ease of use | Between osmotic dilator placement and dilation and evacuation procedure (approximately 16-24 hours)
  Perception of the ease of use of the TENS unit. At the initial 10-minute mark survey, participants will be asked, "How difficult do you feel it will be to use a TENS unit? (0-10 numeric rating scale)". On the final survey (pre-op survey), only participants in the intervention group will be asked, "How difficult was it to use a TENS unit? (0-10 numeric rating scale)". A score of 0 indicates "not difficult at all." A score of 10 indicates "very difficult."
Analgesic use | Between osmotic dilator placement and dilation and evacuation procedure (approximately 16-24 hours)
  Amount of ibuprofen taken and/or other analgesics

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Natavio, MD, MPH, Study Director — Complex Family Planning, The Queens Medical Center, Department of Obstetrics, Gynecology, and Womens Health
Locations (1):
- 1380 Lusitana St. Ste 1004, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: Undecided